CLINICAL TRIAL: NCT04027569
Title: PROMs To Improve Care: A Pragmatic RCT on Standardized and Patient Specific PROMs on Outcomes After Hand Surgery
Brief Title: PROMs To Improve Care- Standardized vs Patient Specific
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics (Research Staffing)
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 52021
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hand Injuries
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PSFS group (Active Comparator): Patients in this arm will complete the patient specific functional scale (PSFS) during their visits
  Interventions: Other: Patient Specific Functional Scale
- PROMIS PF group (Experimental): Patients in this arm will complete the PROMIS Physical Function during their visits
  Interventions: Other: PROMIS PF

INTERVENTIONS:
Other: Patient Specific Functional Scale — A validated patient reported outcome measure that asks patients to write down activities and score them 0 to 10.
  Arms: PSFS group
Other: PROMIS PF — A computer adaptive, validated patient reported outcome measure that measures physical function on a 1 to 100.
  Arms: PROMIS PF group

SUMMARY:
To examine the impact of using 2 validated PROMs during the care of an orthopaedic condition on shared decision making, patient centered care, and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* hand surgery patients over age 18, english fluency and literacy, able to take informed consent

Exclusion Criteria:

-

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2040-11 (Estimated); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) | Immediately after the clinical encounter, same day as clinical encounter
  DCS is a validated tool that measures patient uncertainty about decisions. it is scored 0 to 100, with higher scores indicating greater conflict about the decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Robin N Kamal, MD MBA, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD